CLINICAL TRIAL: NCT05533086
Title: PD-L1 PET Imaging in Patients With the Immunotherapy for Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiaohua Zhu (Other)
Responsible Party: Sponsor-Investigator, Xiaohua Zhu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20220816
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: NSCLC Stage IV; PD-L1 Gene Amplification
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials have shown efficacy of PD1/PD-L1 checkpoint inhibitors in multiple solid tumors, including NSCLC. Whole body information with regard to target presence, drug kinetics and dynamics, as well as binding of PD-L1 targeting agents to the immune system cells is lacking.Molecular imaging of PD-L1 could lead to new insights on heterogeneity of PD-L1 expression in metastatic lesions and be of help in the prediction of response to PD1/PD-L1 inhibitors in a noninvasive manner.

DETAILED DESCRIPTION:
Immunohistochemistry (IHC) is currently the most commonly used method for evaluation of PD-L1 status in cancer patients,including NSCLC. However, biopsies are spatiotemporally limited because of the highly heterogeneous expression of PD-L1. Only 20-40% of PD-L1-positive patients respond to treatment, while 10% of PD-L1-negative patients show a good response to immune checkpoint inhibitors .Patients with false-negative PD-L1 results may miss the chance for targeted therapy.Additionally, the PD-L1 status can change dynamically during the disease process.Therefore, it is necessary to achieve higher response rates, lower toxicity and lower treatment costs by finding assays to better assess PD-L1 expression and screen patients for benefit.

PD-L1 PET imaging provides a new approach to assess PD-L1 expression in NSCLC patients and is expected to overcome the limitations of immunohistochemical ,detection of PD-L1 expression for dynamic visualization in primary and metastatic tumors . First, PET imaging can provide multidimensional three-dimensional data of overall PD-L1 expression in tumors. Second, the whole-body PD-L1 expression level can be assessed, and the heterogeneity of PD-L1 expression between tumors can be studied simultaneously. Third, it is non-invasive and provides information on PD-L1 expression not only before treatment, but also allows monitoring PD-L1 expression several times during treatment ,to screen patients for benefit and guide treatment.

Currently, the FDA-approved 68Ga/68Gagenerator is commercially available, and the cyclotron can produce 68Ga on a large scale. Also, the 68Ga labeling technology is mature. Therefore, 68Ga-PDL1 PET imaging is more easily translatable to the clinical setting. A previous study reported the synthesis and preclinical evaluation of 68Ga-BMS986192, including PD-L1 affinity, metabolic stability, micro PET imaging and in vivo biodistribution in PD-L1 positive and negative transplanted tumors, demonstrating the feasibility of this tracer for in vivo imaging of tumor PD-L1 expression.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subjects must be diagnosed with histologically confirmed stage IV non-small cell lung cancer and >18 years of age with driver mutations (-).

  (2) Planned for anti-PD-1/PD-L1 therapy. (3) At least one easy accessible lesion of which a biopsy can be taken within one month prior to PET scan.

  (4) Subjects must sign informed consent prior to inclusion in this trial.

Exclusion Criteria:

- (1) Female patients during pregnancy and lactation. (2) Patients with psychiatric disease, severe hepatic and renal insufficiency. (3) Patients who refuse anti-PD-1/PD-L1 therapy. (4) Patients who are claustrophobic or unable to undergo PET/CT examination. (5) Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways, except anti-CTLA4 antibody.

(6) Those who, in the opinion of the investigator, are otherwise unsuitable for clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients should be diagnosed with stage IV non-small cell lung cancer. Patients should be eligible for treatment withanti-PD-1/PD-L1 therapy. Patients participating in other trials with this agent may participate in phase one of this study, as long as this does not interfere with either one of the study protocols.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 1 year
  SUVmax

CONTACTS AND LOCATIONS:
Overall Officials: ZHU XIAOHUA, DR, Principal Investigator — Tongji Hospital
Locations (1):
- TongjiHospital, Wuhan, Hubei, China